CLINICAL TRIAL: NCT01789281
Title: An Open-label, Multi-center Everolimus Roll-over Protocol for Patients Who Have Completed a Previous Novartis-sponsored Everolimus Study and Are Judged by the Investigator to Benefit From Continued Everolimus Treatment
Brief Title: Everolimus Roll-over Protocol for Patients Who Have Completed a Previous Novartis-sponsored Everolimus Study.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001C2X01B; 2012-004707-12 (EudraCT Number)
Record Dates: First submitted 2013-02-07; First posted 2013-02-12 (Estimated); Results first posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Neoplasms
Keywords: Neoplasms; Carcinoid tumor; Neuroendocrine tumor
MeSH Terms: conditions — Neoplasms; Carcinoid Tumor; Neuroendocrine Tumors | interventions — Everolimus; Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Everolimus (Experimental): Participants who were receiving everolimus in a Novartis-sponsored study, were not progressing on the current study treatment and were unable to access everolimus treatment outside of a clinical trial. Participants receiving everolimus treatment in combination with Sandostatin LAR Depot on the parent protocol were allowed to continue Sandostatin LAR Depot treatment.
  Interventions: Drug: Everolimus; Drug: Sandostatin LAR Depot

INTERVENTIONS:
Drug: Everolimus — Everolimus was provided by the investigator in 2.5 mg, 5 mg or 10 mg tablets for daily oral administration. The starting dose of everolimus was the same as the last dose that was given in the parent study. Dose modification thereafter was done at the discretion of the Investigator based upon what is in the subject's best interest.
Drug: Sandostatin LAR Depot — Sandostatin LAR Depot was provided by Novartis or by the investigational site considering local regulations. The dose and frequency of Sandostatin LAR Intramuscular injections was the same as the last dose that was given in the parent study.

SUMMARY:
Study to allow access to everolimus for patients who are on everolimus treatment in a Novartis-sponsored study and are benefiting from the treatment as judged by the investigator

DETAILED DESCRIPTION:
This multi-center, open-label roll-over study aimed to better characterize the long-term safety of everolimus in subjects currently being treated in a Novartis-sponsored studies and who were receiving clinical benefit on the current study treatment as judged by the Investigator.

The study was designed to provide continued treatment with everolimus monotherapy to the subjects. Subjects were allowed to continue combination therapy with Sandostatin LAR® Depot if they were receiving this combination therapy on the parent protocol. Subjects were allowed to continue in this roll-over study until they no longer benefitted from the everolimus treatment as judged by the Investigator, discontinued due to toxicities, subject withdrew consent or lost to follow-up, disease progression, protocol non-compliance, or subject death, whichever occurred first. A subject was considered to have reached end of study when everolimus treatment was permanently discontinued.

As per the original protocol, it was designed to collect only serious adverse events (SAEs) and protocol defined adverse events of special interest (AESIs). However, due to the feedback received from health authorities, the protocol was amended in 2016 (3 years after study was initiated) to collect all AEs (non-serious and serious AEs, and AESIs). The protocol was also amended to include an Investigator assessment of clinical benefit at every visit for remaining subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject enrolled in a Novartis-sponsored, CD&MA study receiving everolimus or everolimus plus Sandostatin LAR Depot and fulfilled all their requirements in the parent study
* Subject benefiting from treatment with everolimus, as determined by the guidelines of the parent protocol.

Exclusion Criteria:

* Subject was permanently discontinued from everolimus study treatment in the parent study.
* Subject was receiving everolimus in combination with an unapproved or experimental treatment

Other protocol-defined inclusion/exclusion criteria might apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-05-14 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (22):
- United States (13):
  - Hematology Oncology Services of Arkansas SC, Little Rock, Arkansas
  - Rocky Mountain Cancer Centers SC, Greenwood Village, Colorado
  - Stamford Hospital, Stamford, Connecticut
  - H Lee Moffitt Cancer Center and Research Institute SC-2, Tampa, Florida
  - Central Indiana Cancer Centers SC, Indianapolis, Indiana
  - Crescent City Research Consortium, LLC SC-3, Metairie, Louisiana
  - Mayo Clinic SC-2, Rochester, Minnesota
  - Washington University School of Medicine Dept of Oncology, St Louis, Missouri
  - Nebraska Cancer Specialists Onc Dept, Omaha, Nebraska
  - Clinical Research Alliance, Lake Success, New York
  - New York University Medical Center SC-4, New York, New York
  - Oregon Health and Science University SC-8, Portland, Oregon
  - Utah Cancer Specialists Utah Cancer (2), Salt Lake City, Utah
- Novartis Investigative Site, Prague, Czech Republic, Czechia
- Italy (2):
  - Novartis Investigative Site, Arezzo, AR
  - Novartis Investigative Site, Milan, MI
- Novartis Investigative Site, Groningen, Netherlands
- Novartis Investigative Site, Leningrad Region, Russia, Russia
- Novartis Investigative Site, Seoul, South Korea
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- Novartis Investigative Site, Bangkok, Thailand
- Novartis Investigative Site, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There was no screening period. Patients enrolled into trial directly from the parent protocol.
Groups:
- Everolimus: Participants who were receiving everolimus in a Novartis-sponsored study
- Everolimus+Sandostatin LAR: Participants who were receiving everolimus in combination with Sandostatin LAR depot in a Novartis-sponsored study
Period: Overall Study
Arm/Group | Everolimus | Everolimus+Sandostatin LAR
Started | 22 | 12
Completed | 0 | 2
Not Completed | 22 | 10
Not completed — Disease progression | 15 | 4
Not completed — Adverse Event | 5 | 5
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Administrative problems | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus | Everolimus+Sandostatin LAR | Total
Number analyzed (Participants) | 22 | 12 | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.6 (9.52) | 57.9 (11.30) | 58.4 (10.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 13 | 6 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment. All SAEs were captured in safety database from enrollment. Safety data collection was changed in the protocol amendment released in March 2016: AEs and SAEs were captured in the clinical database from protocol amendment release (18 March 2016). Hence, SAEs from both safety database and clinical database are summarized separately.
Time Frame: SAEs collected in safety database from enrollment to end of treatment (EOT) plus 30 days, up to approximately 7.2 years. AEs/SAEs collected in clinical database from protocol amendment date 18 March 2016 to EOT plus 30 days, up to approximately 4.5 years
Population: All subjects who received at least one dose of everolimus after enrolling into the roll-over study.
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus | Everolimus+Sandostatin LAR
Number analyzed (Participants) | 22 | 12
Participants
  SAEs (Safety database) | 6 | 9
  Treatment-related SAEs (Safety database) | 1 | 4
  AEs (Clinical Database) | 7 | 7
  Tretament-related AEs (Clinical Database) | 4 | 4
  SAEs (Clinical Database) | 2 | 4
  Treatment-related SAEs (Clinical Database) | 0 | 2

2. Secondary Outcome: Percentage of Patients With Clinical Benefit
Description: Percentage of patients with clinical benefit as judged by the investigator. Investigator attestation of continued clinical benefit was collected in clinical database after protocol amendment (release date 18 March 2016). Clinical benefit assessment before protocol amendment was done retrospectively.
Time Frame: After 3 months from enrollment, every 3 months, until end of treatment, assessed up to 7.2 years
Population: All participants who remained in the study after protocol amendment (18 March 2016) with at least one assessment reported for the specified endpoint
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus | Everolimus+Sandostatin LAR
Number analyzed (Participants) | 9 | 7
Participants
  At 3 months | 9 | 7
  At 6 months | 8 | 7
  At 9 months | 8 | 7
  At 12 months | 8 | 7
  At 15 months | 8 | 7
  At 18 months | 8 | 7
  At 21 months | 8 | 7
  At 24 months | 6 | 7
  At 27 months | 5 | 7
  At 30 months | 3 | 7
  At 33 months | 2 | 7
  At 36 months | 1 | 7
  At 39 months | 1 | 7
  At 42 months | 1 | 6
  At 45 months | 1 | 6
  At 48 months | 1 | 6
  At 51 months | 1 | 6
  At 54 months | 0 | 6
  At 57 months | 0 | 5
  At 60 months | 0 | 5
  At 63 months | 0 | 4
  At 66 months | 0 | 4
  At 69 months | 0 | 3
  At 72 months | 0 | 3
  At 75 months | 0 | 3
  At 78 months | 0 | 2
  At 81 months | 0 | 1
  At 84 months | 0 | 0

ADVERSE EVENTS:
Time Frame: SAEs were collected in safety database from enrollment to end of the treatment (EOT) plus 30 days, up to approximately 7.2 years. Other AEs (Non-serious AEs) were collected in clinical database from protocol amendment date 18 March 2016 to EOT plus 30 days, up to approximately 4.5 years
Description: Any sign or symptom that occurs during the study treatment plus 30 days post treatment. SAEs were collected throughout the study duration in the safety database. Other AEs (Non-serious AEs) were collected after global protocol amendment date 18-Mar-2016 in the clinical database.
Groups:
- Everolimus + Sandostatin LAR: Participants who were receiving everolimus in combination with Sandostatin LAR depot in a Novartis-sponsored study
- All Subjects: All subjects
Arm/Group | Everolimus | Everolimus + Sandostatin LAR | All Subjects
All-Cause Mortality (participants affected / at risk) | 1/22 | 2/12 | 3/34
Serious Adverse Events (participants affected / at risk) | 6/22 | 9/12 | 15/34
Other Adverse Events (participants affected / at risk) | 3/22 | 5/12 | 8/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=22) | Everolimus + Sandostatin LAR (N=12) | All Subjects (N=34)
Aplastic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 2 | 2
Heart valve incompetence (Cardiac disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 1
Asthenia (General disorders) | 0 | 1 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 2 | 3 | 5
Pyelonephritis (Infections and infestations) | 0 | 1 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 1
Fluid intake reduced (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 2
Nephropathy (Renal and urinary disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1
Haemorrhage (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=22) | Everolimus + Sandostatin LAR (N=12) | All Subjects (N=34)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1 | 1
Periorbital oedema (Eye disorders) | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Duodenal stenosis (Gastrointestinal disorders) | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2 | 2
Fatigue (General disorders) | 1 | 1 | 2
Oedema peripheral (General disorders) | 0 | 2 | 2
Pain (General disorders) | 0 | 1 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Blood chromogranin A increased (Investigations) | 0 | 1 | 1
Blood triglycerides increased (Investigations) | 0 | 1 | 1
Weight decreased (Investigations) | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 2 | 2
Depression (Psychiatric disorders) | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
The original protocol was designed to collect only SAEs and protocol defined AESIs in the Safety database. The protocol was amended in 2016 (3 years after study was initiated) to include all AEs (non-SAEs, SAEs, and AESIs) to be collected in the clinical database. At the time of amendment release, 32 of the 34 subjects were enrolled and did not have AEs collected in clinical database before protocol amendment, which also amounts to approximately 50% of SAEs not reported in clinical database.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-03-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT01789281/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/81/NCT01789281/SAP_001.pdf